CLINICAL TRIAL: NCT03383783
Title: Evaluation of the Fluoride Dose Response of a Modified In Situ Caries Model
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Domenick Zero (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Domenick Zero, Director, Oral Health Research Institute, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 17-I-112; 208705 (Other: GlaxoSmithKline)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Caries
Keywords: Caries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment Period 1 (Other): 0 ppm F (placebo, negative control), 250 ppm F as NaF (dose-response control), 500 ppm F as NaF (dose-response control), 1100 ppm F as NaF (positive control)
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 250 ppm F as NaF (dose-response control); Drug: 500 ppm F as NaF (dose-response control); Drug: 1100 ppm F as NaF (positive control)
- Treatment Period 2 (Other): 0 ppm F (placebo, negative control), 250 ppm F as NaF (dose-response control), 500 ppm F as NaF (dose-response control), 1100 ppm F as NaF (positive control)
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 250 ppm F as NaF (dose-response control); Drug: 500 ppm F as NaF (dose-response control); Drug: 1100 ppm F as NaF (positive control)
- Treatment Period 3 (Other): 0 ppm F (placebo, negative control), 250 ppm F as NaF (dose-response control), 500 ppm F as NaF (dose-response control), 1100 ppm F as NaF (positive control)
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 250 ppm F as NaF (dose-response control); Drug: 500 ppm F as NaF (dose-response control); Drug: 1100 ppm F as NaF (positive control)
- Treatment Period 4 (Other): 0 ppm F (placebo, negative control), 250 ppm F as NaF (dose-response control), 500 ppm F as NaF (dose-response control), 1100 ppm F as NaF (positive control)
  Interventions: Drug: 0 ppm F (placebo, negative control); Drug: 250 ppm F as NaF (dose-response control); Drug: 500 ppm F as NaF (dose-response control); Drug: 1100 ppm F as NaF (positive control)

INTERVENTIONS:
Drug: 0 ppm F (placebo, negative control) — Each subject will use this product during one of the four treatment periods in the crossover study design.
  Other Names: Sensodyne sodium fluoride/silica toothpaste base formulation
Drug: 250 ppm F as NaF (dose-response control) — Each subject will use this product during one of the four treatment periods in the crossover study design.
  Other Names: Sensodyne sodium fluoride/silica toothpaste base formulation
Drug: 500 ppm F as NaF (dose-response control) — Each subject will use this product during one of the four treatment periods in the crossover study design.
  Other Names: Sensodyne sodium fluoride/silica toothpaste base formulation
Drug: 1100 ppm F as NaF (positive control) — Each subject will use this product during one of the four treatment periods in the crossover study design.
  Other Names: Sensodyne sodium fluoride/silica toothpaste base formulation

SUMMARY:
The purpose of this study is to evaluate the fluoride dose response of different dentifrice fluoride concentrations - 0, 250, 500 and 1100 ppm fluoride of our existing in situ model involving the use of human enamel specimens placed in the buccal flange area of the subjects partial denture with the modified model involving placement of bovine enamel specimens in a denture tooth location.

DETAILED DESCRIPTION:
This will be a double blind, single center, 4-way crossover design study involving 34 adult subjects, between the ages of 18 and 85 years. Two to three days before the start of each treatment period the subjects will have their teeth cleaned to remove all accessible plaque and calculus and will be provided with a non-fluoride dentifrice to use until their next visit. At the beginning of each testing period, two gauze-covered 4 × 4 mm partially demineralized human enamel specimens will be placed in the buccal flange area of the subject's mandibular partial denture. In addition, two gauze-covered 4 mm round partially demineralized bovine enamel specimens will be placed in the buccal surface of two posterior denture teeth of the same side of the partial denture. Once specimens are placed, subjects will wear their partial dentures twenty-four hours a day and use their assigned toothpaste twice daily, as instructed, until their next visit. Specimens will be removed after two weeks and the subjects will undergo a four to five day washout period followed by another cleaning and two to three day lead in period. This process will be repeated until all subjects have used all four test products. Changes in the mineral content of the enamel specimens will be assessed using the SMH and TMR. Enamel fluoride uptake (EFU) will be determined using the microdrill enamel biopsy technique. In addition the net acid resistance (NAR) and the comparative acid resistance (CAR) of the remineralized enamel specimens will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. provide voluntary, written informed consent;
2. be between 18 and 85 years old;
3. understand and be willing, able and likely to comply with all study procedures and restrictions;
4. be wearing a removable mandibular partial denture with sufficient room in one posterior buccal flange area to accommodate two enamel specimens (required dimensions 12 × 7 mm) and room on the same side to accommodate two 4 mm round specimens in the buccal surface of two posterior denture teeth;
5. be willing and capable of wearing their removable partial denture 24 hours a day for four (4), two-week treatment periods;
6. be willing to allow study personnel to drill specimen sites (as described #4) in their mandibular partial denture;
7. be in good medical and dental health with no active caries or periodontal disease; NOTE; subjects presenting at screening with caries may continue in the study if their carious lesions are restored prior to beginning treatment 1.
8. have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate ≥ 0.2 mL/min; gum base stimulated whole saliva flow rate ≥ 0.8 mL/min).

Exclusion Criteria:

1. currently be pregnant, intending to become pregnant during the study period or breast feeding;
2. currently have any medical condition that could be expected to interfere with the subject's safety during the study period;
3. currently be taking antibiotics or have taken antibiotics in the two weeks prior to the beginning treatment 1;
4. have participated in another clinical study or receipt of an investigational drug within 30 days of beginning treatment 1; or
5. be taking fluoride supplements, required to use a fluoride mouthrinse or have received a professional fluoride treatment in the two weeks preceding specimen placement;
6. be taking or have ever taken bisphosphonate drugs (e.g., Fosamax, Actonel and Boniva) for the treatment of osteoporosis;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domenick T Zero, DDS, MS, Principal Investigator — Indiana University; Anderson Hara, DDS, PhD, Principal Investigator — Indiana University; Frank Lippert, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Dentistry, Oral Health Research Institute, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant signed the informed consent and attended up to visit 2, but were dropped from the study as they no longer met inclusion criteria, and this occurred before randomization to interventions.
Groups:
- All Study Participants: This was a 4-way crossover design study. All participants were randomized to receive the following interventions:
  Dentifrice fluoride concentrations - 0, 250, 500 and 1100 ppm fluoride of our existing in situ model involving the use of human enamel specimens placed in the buccal flange area of the subjects partial denture with the modified model involving placement of bovine enamel specimens in a denture tooth location.
Period: Overall Study
Arm/Group | All Study Participants
Started | 27
Completed | 25
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Full Range); unit: Years] | 67 [37 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  White/African-American | 1
  African-American | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Microhardness Recovery (%SMH)
Description: The extent of remineralization will be calculated based on the method of [Gelhard et al., 1979].
  * SMH recovery = (D1-R)/(D1-B) ×100 B = indentation length (µm) of sound enamel specimen at baseline D1 = indentation length (µm) after in vitro demineralization R = indentation length (µm) after intra-oral exposure.
Time Frame: Enamel specimens will be evaluated after 14 days of intra-oral exposure
Measure: Mean (95% Confidence Interval); unit: Percent Surface Microhardness Recovery
Groups:
- Bovine Specimens 0 Ppm F: This arm group consisted of the two bovine specimens and 0 parts per million fluoride dentifrice.
- Bovine Specimens 250 Ppm F: This arm group consisted of the two bovine specimens and 250 parts per million fluoride dentifrice.
- Bovine Specimens 500 Ppm F: This arm group consisted of the two bovine specimens and 500 parts per million fluoride dentifrice.
- Bovine Specimens 1100 Ppm F: This arm group consisted of the two bovine specimens and 1100 parts per million fluoride dentifrice.
- Human Specimens 0 Ppm F: This arm group consisted of the two human specimens and 0 parts per million fluoride dentifrice.
- Human Specimens 250 Ppm F: This arm group consisted of the two human specimens and 250 parts per million fluoride dentifrice.
- Human Specimens 500 Ppm F: This arm group consisted of the two human specimens and 500 parts per million fluoride dentifrice.
- Human Specimens 1100 Ppm F: This arm group consisted of the two human specimens and 1100 parts per million fluoride dentifrice.
Arm/Group | Bovine Specimens 0 Ppm F | Bovine Specimens 250 Ppm F | Bovine Specimens 500 Ppm F | Bovine Specimens 1100 Ppm F | Human Specimens 0 Ppm F | Human Specimens 250 Ppm F | Human Specimens 500 Ppm F | Human Specimens 1100 Ppm F
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
Percent Surface Microhardness Recovery | 13.96 [8 to 20.29] | 30.59 [22.26 to 38.71] | 40.74 [31.68 to 50.34] | 48.28 [37.15 to 57.86] | 7.42 [2.55 to 12.45] | 16.27 [10.33 to 22.51] | 21.59 [13.67 to 29.64] | 26.75 [18.19 to 35.29]

2. Secondary Outcome: Net Acid Resistance (NAR)
Description: The %NAR will be calculated by the method of Corpron [Corpron et al., 1986]:
  * Net Acid Resistance = [(D1-D2) / (D1-B)] * 100 B= Indentation length (µm) of sound enamel at baseline D1= Indentation length (µm) after first in vitro demineralization D2= Indentation length (µm) after second in vitro demineralization
Time Frame: Enamel specimens will be evaluated after 14 days of intra-oral exposure
Measure: Mean (95% Confidence Interval); unit: % Net Acid Resistance
Arm/Group | Bovine Specimens 0 Ppm F | Bovine Specimens 250 Ppm F | Bovine Specimens 500 Ppm F | Bovine Specimens 1100 Ppm F | Human Specimens 0 Ppm F | Human Specimens 250 Ppm F | Human Specimens 500 Ppm F | Human Specimens 1100 Ppm F
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
% Net Acid Resistance | -22.68 [-36.71 to -11.7] | 11.43 [1.92 to 20.42] | 18.66 [8.17 to 27.63] | 31.79 [17.57 to 42.9] | -18.60 [-28.62 to -9.55] | 1.99 [-6.31 to 9.43] | 8.31 [-1.36 to 16.9] | 16.87 [8.91 to 23.95]

3. Secondary Outcome: Comparative Acid Resistance (CAR)
Description: Using the data from the four centrally located enamel specimens, the equation used will compare explicitly the reduction in SMH brought by the first and second acid challenges:
  * Comparative Acid Resistance = [(D2-R) / (D1-B)] * 100 B= Indentation length (µm) of sound enamel at baseline R= Indentation length (µm) of enamel after in situ remineralization D1= Indentation length (µm) after first in vitro demineralization D2= Indentation length (µm) after second in vitro demineralization
Time Frame: Enamel specimens will be evaluated after 14 days of intra-oral exposure
Measure: Mean (95% Confidence Interval); unit: % Comparative Acid Resistance
Arm/Group | Bovine Specimens 0 Ppm F | Bovine Specimens 250 Ppm F | Bovine Specimens 500 Ppm F | Bovine Specimens 1100 Ppm F | Human Specimens 0 Ppm F | Human Specimens 250 Ppm F | Human Specimens 500 Ppm F | Human Specimens 1100 Ppm F
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
% Comparative Acid Resistance | 36.42 [23.87 to 51.03] | 19.20 [11.28 to 27.99] | 22.16 [13 to 32.82] | 16.27 [8.98 to 24.46] | 25.82 [18.14 to 33.79] | 14.31 [9.74 to 19.53] | 13.33 [8.59 to 18.82] | 9.71 [4.98 to 14.53]

4. Secondary Outcome: Enamel Fluoride Uptake (EFU)
Description: The amount of fluoride-uptake by enamel will be calculated based on the amount of fluoride divided by the area of the enamel cores and expressed as µg F/cm2.
Time Frame: Enamel specimens will be evaluated after 14 days of intra-oral exposure
Measure: Mean (95% Confidence Interval); unit: µg F/cm^2
Arm/Group | Bovine Specimens 0 Ppm F | Bovine Specimens 250 Ppm F | Bovine Specimens 500 Ppm F | Bovine Specimens 1100 Ppm F | Human Specimens 0 Ppm F | Human Specimens 250 Ppm F | Human Specimens 500 Ppm F | Human Specimens 1100 Ppm F
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
µg F/cm^2 | 0.96 [0.73 to 1.16] | 2.25 [1.94 to 2.56] | 2.69 [2.35 to 2.97] | 2.98 [2.62 to 3.27] | 0.96 [0.77 to 1.15] | 2.14 [1.9 to 2.38] | 2.50 [2.32 to 2.71] | 2.73 [2.48 to 2.94]

5. Secondary Outcome: Transverse Microradiography (TMR) - Integrated Mineral Loss - ∆Z
Description: Lesions will be analyzed after in situ demineralization and the following three parameters calculated:
  1. Integrated Mineral Loss - ∆Z= [(lesion depth x 87) - area under the curve*]
  2. Lesion Depth - L (83% mineral i.e. 95% of the mineral content of sound enamel)
  3. Maximum mineral density at the surface-zone - SZmax
Time Frame: Enamel specimens will be evaluated after 14 days of intra-oral exposure
Measure: Mean (95% Confidence Interval); unit: Integrated Mineral Loss - ∆Z
Arm/Group | Bovine Specimens 0 Ppm F | Bovine Specimens 250 Ppm F | Bovine Specimens 500 Ppm F | Bovine Specimens 1100 Ppm F | Human Specimens 0 Ppm F | Human Specimens 250 Ppm F | Human Specimens 500 Ppm F | Human Specimens 1100 Ppm F
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
Integrated Mineral Loss - ∆Z | 1240 [948 to 1621] | 902 [710 to 1136] | 664 [546 to 803] | 684 [552 to 841] | 1526 [1250 to 1832] | 912 [793 to 1033] | 901 [800 to 1019] | 859 [754 to 966]

6. Secondary Outcome: Transverse Microradiography (TMR) - Lesion Depth - L
Description: as for outcome 5
Time Frame: Enamel specimens will be evaluated after 14 days of intra-oral exposure
Measure: Mean (95% Confidence Interval); unit: Micrometers
Arm/Group | Bovine Specimens 0 Ppm F | Bovine Specimens 250 Ppm F | Bovine Specimens 500 Ppm F | Bovine Specimens 1100 Ppm F | Human Specimens 0 Ppm F | Human Specimens 250 Ppm F | Human Specimens 500 Ppm F | Human Specimens 1100 Ppm F
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
Micrometers | 52.01 [40.62 to 65.49] | 41.74 [32.58 to 53.38] | 34.85 [27.39 to 43.65] | 27.31 [22.62 to 32.18] | 60.73 [50.56 to 71.99] | 42.12 [34.28 to 49.8] | 37.38 [31.17 to 45.06] | 36.02 [31.03 to 41.21]

7. Secondary Outcome: Transverse Microradiography (TMR) - Maximum Mineral Density at the Surface-zone
Description: Lesions will be analyzed after in situ demineralization and the following three parameters calculated:
  1. Integrated Mineral Loss - ∆Z= [(lesion depth x 87) - area under the curve*]
  2. Lesion Depth - L (83% mineral i.e. 95% of the mineral content of sound enamel)
  3. Maximum mineral density at the surface-zone - SZmax (arbitrary unit from TMR software)
Time Frame: Enamel specimens will be evaluated after 14 days of intra-oral exposure
Measure: Mean (95% Confidence Interval); unit: SZmax
Arm/Group | Bovine Specimens 0 Ppm F | Bovine Specimens 250 Ppm F | Bovine Specimens 500 Ppm F | Bovine Specimens 1100 Ppm F | Human Specimens 0 Ppm F | Human Specimens 250 Ppm F | Human Specimens 500 Ppm F | Human Specimens 1100 Ppm F
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
SZmax | 62.17 [59.59 to 64.44] | 62.54 [60.14 to 65.14] | 67.13 [63.53 to 70.61] | 65.93 [60.31 to 70.88] | 61.22 [58.82 to 63.62] | 62.99 [60.59 to 65.42] | 61.38 [59.32 to 63.24] | 63.66 [61.14 to 66.47]

ADVERSE EVENTS:
Time Frame: Each participant was monitored for a 3 month period.
Description: The collection/monitoring of adverse events started at visit 2 (prior to randomization), at which time there were 28 eligible subjects. Human and bovine specimens were both placed on the same side of the lower partial dentures in 27 subjects at visit 3 (randomization), and from that point forward adverse events were monitored based on the assigned treatment.
Groups:
- 0 Ppm F: 0 parts per million fluoride
- 250 Ppm F: 250 parts per million fluoride
- 500 Ppm F: 500 parts per million fluoride
- 1100 Ppm F: 1100 parts per million fluoride
- Between Treatment Periods: Adverse Events that occurred between treatment periods.
- Prior to Randomization: Adverse Events that occurred prior to a subject being randomized into the study.
Arm/Group | 0 Ppm F | 250 Ppm F | 500 Ppm F | 1100 Ppm F | Between Treatment Periods | Prior to Randomization
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 10/27 | 5/27 | 6/27 | 5/27 | 7/27 | 18/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0 Ppm F (N=27) | 250 Ppm F (N=27) | 500 Ppm F (N=27) | 1100 Ppm F (N=27) | Between Treatment Periods (N=27) | Prior to Randomization (N=28)
Mouth Erythema (Gastrointestinal disorders) | 1 (1) | 2 (3) | 4 (4) | 3 (4) | 0 (0) | 5 (5)
Back Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Common Cold (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enlarged Lymphnode (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gum Tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected Cysts (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leg Cramps (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loose Crown (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lost Filling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 2 (2) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal White Patch (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Stiffness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Epitaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Burning Sensation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Shoulder Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Headache (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen Eye Lid (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth Extraction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT03383783/Prot_SAP_000.pdf